CLINICAL TRIAL: NCT00738062
Title: An Open-label Study, to Assess the Long-term Safety and Clinical Benefit of Droxidopa in Subjects With PAF, Dopamine Beta Hydroxylase Deficiency or Non-diabetic Neuropathy and Symptomatic Neurogenic Orthostatic Hypotension
Brief Title: Open-Label Clinical Study of Droxidopa in Patients With Neurogenic Orthostatic Hypotension (NOH)
Acronym: NOH303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Droxidopa NOH303
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Neurogenic Orthostatic Hypotension; Non-Diabetic Autonomic Neuropathy; Multiple System Atrophy; Dopamine Beta Hydroxylase Deficiency
Keywords: NOH; Neurogenic Orthostatic Hypotension; Orthostatic hypotension; PAF; Pure Autonomic Failure; MSA; Multiple System Atrophy; Neuropathy; Autonomic Failure; Parkinson; Dopamine Deficiency; Dopamine; Droxidopa
MeSH Terms: conditions — Multiple System Atrophy; dopamine beta hydroxylase deficiency; Hypotension, Orthostatic; Pure Autonomic Failure | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Droxidopa (Active Comparator): Study medication
  Interventions: Drug: Droxidopa
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Droxidopa — 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
  Arms: Droxidopa
Drug: Placebo — 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
  Other Names: Inactive drug (to look like Droxidopa)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the durability of effect of Droxidopa in treating symptoms of neurogenic orthostatic hypotension in patients with Primary Autonomic Failure (Pure Autonomic Failure, Multiple System Atrophy, Parkinson's Disease), Non-diabetic neuropathy, or Beta Hydroxylase deficiency.

DETAILED DESCRIPTION:
Systolic blood pressure is transiently and minimally decreased in healthy individuals upon standing. Normal physiologic feedback mechanisms work through neurally-mediated pathways to maintain the standing blood pressure, and thus maintain adequate cerebral perfusion. The compensatory mechanisms that regulate blood pressure upon standing are dysfunctional in subjects with orthostatic hypotension (OH), a condition that may lead to inadequate cerebral perfusion with accompanying symptoms of syncope, dizziness or lightheadedness, unsteadiness and blurred or impaired vision, among other symptoms.

The autonomic nervous system has a central role in the regulation of blood pressure. Primary Autonomic Failure is manifested in a variety of syndromes. Orthostatic hypotension is a usual presenting symptom. Primary Autonomic Failure may be the primary diagnosis, and classifications include pure autonomic failure (PAF), also called idiopathic orthostatic hypotension (Bradbury-Eggleston syndrome) autonomic failure with multiple system atrophy (Shy-Drager syndrome) and also Parkinson's disease. Regardless of the primary condition, autonomic dysfunction underlies orthostatic hypotension.

Orthostatic hypotension may be a severely disabling condition which can seriously interfere with the quality of life of afflicted subjects. Currently available therapeutic options provide some symptomatic relief in a subset of subjects, but are relatively ineffective and are often accompanied by severe side effects that limit their usefulness. Support garments (tight-fitting leotard) may prove useful in some subjects, but is difficult to don without family or nursing assistance, especially for older subjects. Midodrine, fludrocortisone, methylphenidate, ephedrine, indomethacin and dihydroergotamine are among some of the pharmacological interventions that have been used to treat orthostatic hypotension, although only midodrine is specifically approved for this indication. The limitations of these currently available therapeutic options, and the incapacitating nature and often progressive downhill course of disease, point to the need for an improved therapeutic alternative.

The current withdrawal design study will measure the efficacy of droxidopa on symptoms of neurogenic orthostatic hypotension in patients randomized to continued droxidopa treatment versus placebo, following 14 days of double-blind treatment.

Droxidopa

Droxidopa [also, known as L-threo-3,4-dihydroxyphenylserine, L-threo-DOPS, or L-DOPS] is the International non-proprietary name (INN) for a synthetic amino acid precursor of norepinephrine (NE), which was originally developed by Sumitomo Pharmaceuticals Co., Limited, Japan. It has been approved for use in Japan since 1989. Droxidopa has been shown to improve symptoms of orthostatic hypotension that result from a variety of conditions including Shy Drager syndrome (Multiple System Atrophy), Pure Autonomic Failure, and Parkinson's disease. There are four stereoisomers of DOPS; however, only the L-threo-enantiomer (droxidopa) is biologically active.

The exact mechanism of action of droxidopa in the treatment of symptomatic NOH has not been precisely defined; however, its NE replenishing properties with concomitant recovery of decreased noradrenergic activity are considered to be of major importance.

Droxidopa has been marketed in Japan since 1989. Data from clinical studies and post-marketing surveillance programs conducted in Japan show that the most commonly reported adverse drug reactions with droxidopa are increased blood pressure, nausea, and headache. In clinical studies, the prevalence and severity of droxidopa adverse effects appear to be similar to those reported by the placebo control arm.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, each patient must fulfill the following criteria:

* Participated in Droxidopa Protocol 302;
* Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care.

Exclusion Criteria:

Patients are not eligible for this study if they fulfill one or more of the following criteria:

* Currently taking ephedrine or midodrine;
* Patients taking ephedrine or midodrine must stop taking these drugs at least 2 days prior to their study entry visit (Visit 1).
* Currently taking anti-hypertensive medication;

  * The use of short-acting anti-hypertensive medications at bedtime is permitted.
* Currently taking tri-cyclic antidepressant medication or other norepinephrine re-uptake inhibitors;
* Have changed dose, frequency and or type of prescribed medication, within two weeks of study start (excluding ephedrine and midodrine);
* History of more than moderate alcohol consumption;
* History of known or suspected drug or substance abuse;
* Women of childbearing potential who are not using a medically accepted contraception;

  * Reproductive potential:
  * Female subjects should be either post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile, or women of child-bearing potential (WOCP) who are using or agree to use acceptable methods of contraception.
  * Acceptable contraceptives include intrauterine devices (IUDs), hormonal contraceptives (oral, depot, patch or injectable) and double barrier methods such as condoms or diaphragms with spermicidal gel or foam.
  * For WOCP a urine pregnancy test must be conducted at each study visit.
  * WOCP must be advised to use acceptable contraceptives throughout the study period and for 30 days after the last dose of investigational product.
  * If hormonal contraceptives are used they should be taken according to the package insert.
  * WOCP who are not currently sexually active must agree to use acceptable contraception, as defined above, if they decide to become sexually active during the period of the study and for 30 days after the last dose of investigational product.
* Sexually active males whose partner is a WOCP and who do not agree to use condoms for the duration of the study and for 30 days after the last dose;
* Women who are pregnant or breast feeding;
* Known or suspected hypersensitivity to the study medication or any of its ingredients;
* Pre-existing sustained severe hypertension (BP 180/110 mmHg in the sitting position);
* Have atrial fibrillation or, in the investigator's opinion, have any other significant cardiac arrhythmia;
* Any other significant systemic, hepatic, cardiac or renal illness;
* Diabetes mellitus or insipidus;
* Have a history of closed angle glaucoma;
* Have a known or suspected malignancy;
* Have a serum creatinine level > 130 umol/L;
* Patients with known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug;
* In the investigator's opinion, have clinically significant abnormalities on clinical examination or laboratory testing;
* In the investigator's opinion, are unable to adequately co-operate because of individual or family situation;
* In the investigator's opinion, are suffering from a mental disorder that interferes with the diagnosis and/or with the conduct of the study, e.g. schizophrenia, major depression, dementia;
* Are not able or willing to comply with the study requirements for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann Kaufmann, MD, Principal Investigator — NYU School of Medicine; Christopher J. Mathias, MD, Principal Investigator — Imperial School of Medicine
Locations (54):
- United States (44):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dedicated Clinical Research, Litchfield Park, Arizona
  - Xenoscience Inc., Phoenix, Arizona
  - Sun Health Research Institute, Sun City, Arizona
  - The Parkinson's and Movement Disorders Institute, Fountain Valley, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - The Parkinson's Institute, Sunnyvale, California
  - Electrophysiology Associates, Colorado Springs, Colorado
  - Parkinson's Disease & Movment Disorder Center, Boca Raton, Florida
  - Southeastern Integrated Medical, Gainesville, Florida
  - Mayo Jacksonville Florida Department of Neurology, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Medical Associates of North Georgia, Canton, Georgia
  - Saint Mary of Nazareth Hospital Center, Chicago, Illinois
  - North Chicago VA Medical Center, North Chicago, Illinois
  - Indiana Medical Research, Elkhart, Indiana
  - JWM Neurology, Indianapolis, Indiana
  - Kansas City Bone and Joint, PA, Overland Park, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Henry Ford Health System, Southfield, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - New Jersey Neuroscience Institute, Edison, New Jersey
  - Kingston Neurological Associates, PC, Kingston, New York
  - NYU Medical Center, New York, New York
  - Columbia University Neurological institute of NY, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Jacinto Medical Group, PA, Baytown, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Scott & White Healthcare - Round Rock, Round Rock, Texas
  - Scott & White Memorial Hospital & Clinic, Temple, Texas
  - East Texas Medical Center - Neurological Institute Movment Disorders Center, Tyler, Texas
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Baker Heart Research Institute, Melbourne, Victoria
  - Austin Hospital, Heidelburg
- Canada (5):
  - McMaster University, Hamilton, Ontario
  - Centre for Movement Disorders, Markham, Ontario
  - Parkinson's & Neurodegenerative Disorders Clinic, Ottawa, Ontario
  - SMBD Jewish General Hospital - Department of Neurology, Montreal, Quebec
  - Quebec Memory and Motor Skills Disorders Clinic, Québec, Quebec
- New Zealand (2):
  - Auckland Hospital, Grafton Auckland, Private Bag
  - Van der Veer Institute for Parkinson's Disease and Movement Disorders, Christchurch

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Droxidopa: 3 months of open-label treatment with droxidopa (t.i.d., at optimal dose)
- Double-blind Droxidopa: Double-blind
  Droxidopa: 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
- Double-blind Placebo: Double-blind
  Placebo: 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
Period: Open Label Treatment
Arm/Group | Open-Label Droxidopa | Double-blind Droxidopa | Double-blind Placebo
Started | 103 | 0 | 0
Completed | 75 | 0 | 0
Not Completed | 28 | 0 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0
Not completed — Adverse Event | 11 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Investigator Decision | 1 | 0 | 0
Period: 2 Week Randomized Withdrawal
Arm/Group | Open-Label Droxidopa | Double-blind Droxidopa | Double-blind Placebo
Started | 0 (Patients completing the open label titration phase were randomized to either Droxidopa or Placebo) | 38 | 37
Completed | 0 | 38 | 37
Not Completed | 0 | 0 | 0
Period: Open-Label Extension
Arm/Group | Open-Label Droxidopa | Double-blind Droxidopa | Double-blind Placebo
Started | 74 (One patient completed double blind randomization but did not enter the open label extension) | 0 | 0
Completed | 57 | 0 | 0
Not Completed | 17 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Study Terminated | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Omits 1 patient who randomized into the study in error and did not receive study drug.
Groups:
- Open-Label Droxidopa: Only participated in 3 months of open-label treatment with droxidopa (t.i.d., at optimal dose)
- Total: Total of all reporting groups
Arm/Group | Open-Label Droxidopa | Double-blind Droxidopa | Double-blind Placebo | Total
Number analyzed (Participants) | 27 | 38 | 37 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10.95) | 68.2 (13.03) | 66.2 (12.09) | 65.8 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 13 | 41
  Male | 14 | 23 | 24 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 27 | 37 | 36 | 100
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 25 | 22 | 63
  Canada | 2 | 6 | 3 | 11
  Australia | 2 | 2 | 2 | 6
  New Zealand | 0 | 1 | 1 | 2
  United Kingdom | 0 | 1 | 3 | 4
  Poland | 7 | 3 | 6 | 16
Primary Clinical Diagnosis [Number; unit: participants]
  Parkinson's Disease | 10 | 20 | 18 | 48
  Multiple System Atrophy | 10 | 8 | 9 | 27
  Pure Autonomic Failure | 3 | 8 | 7 | 18
  Dopamine Beta-Hydroxylase Deficiency | 0 | 1 | 0 | 1
  Non-Diabetic Autonomic Neuropathy | 3 | 0 | 2 | 5
  Other | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Orthostatic Hypotension Questionnaire Composite Score (OHQ)
Description: The OHQ is the average of two sub-scales, the Orthostatic Hypotension Symptom Assessment Scale (OHSA) and the Orthostatic Hypotension Daily Activities Scale (OHDAS). Each asks the patient to rate their symptoms or disease impact over the past week. The OHSA sub-scale is the average of six items: 1) Dizziness, lightheadedness, feeling faint or feeling like you might black out; 2) Problems with vision; 3) Weakness; 4) Fatigue; 5) Trouble concentrating; and 6) Head/neck discomfort. The OHDAS sub-scale is the average of four items: 1) Standing for a short time; 2) Standing for a long time; 3) Walking for a short time; and 4) Walking for a long time. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe.
  In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug). All patients are on open-label droxidopa for 3 months prior to randomization.
Time Frame: 14 days
Population: The analysis population was based on the ITT population of all patients randomized. Last observation carry forward was used for patients who prematurely discontinued the study.
  One droxidopa patient was excluded from the analysis because OHQ values were not evaluable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 37 | 37
units on a scale | 0.57 (1.891) | 0.90 (1.550)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.438, Mantel Haenszel; Mantel-Haenszel statistic comparing treatment groups based on rank statistics adjusted for the covariate OHSA Item 1 value at randomization

2. Secondary Outcome: Change in Orthostatic Hypotension Daily Activities (OHDAS) Score
Description: The OHDAS scale is the average of four items: 1) Standing for a short time; 2) Standing for a long time; 3) Walking for a short time; and 4) Walking for a long time. Each asks the patient to rate their disease impact over the past week. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe.
  Change: score at end of randomization minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug).
Time Frame: 14 days
Population: One droxidopa patient excluded from analysis because data were not evaluable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 37 | 37
units on a scale | 0.53 (2.204) | 0.71 (1.629)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.554, Mantel Haenszel; Mantel-Haenszel statistic comparing treatment groups based on rank statistics adjusted for the covariate OHDAS Composite value at randomization

3. Secondary Outcome: Change in Orthostatic Hypotension Symptom Assessment (OHSA) Composite Score
Description: The OHSA scale is the average of six items: 1) Dizziness, lightheadedness, feeling faint or feeling like you might black out; 2) Problems with vision; 3) Weakness; 4) Fatigue; 5) Trouble concentrating; and 6) Head/neck discomfort. Each asks the patient to rate their symptoms over the past week. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe.
  Change: score at end of randomization minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 38 | 37
units on a scale | 0.59 (1.963) | 1.10 (1.658)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.198, Mantel Haenszel; Mantel-Haenszel statistic comparing treatment groups based on rank statistics adjusted for the covariate OHSA Composite value at baseline

4. Secondary Outcome: Change in Systolic Blood Pressure (SBP) Measurements 3 Minutes Post Standing
Description: Change: standing systolic blood pressure at end of study minus standing systolic blood pressure at randomization. In this withdrawal design, a negative score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug). All patients are on open-label droxidopa for 3 months prior to randomization to either continued droxidopa or to placebo.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 38 | 37
mmHg | -8.4 (26.63) | 0.0 (18.51)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.286, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]

5. Post Hoc Outcome: Change in Dizziness/ Lightheadedness/ Feeling Faint/ or Feeling Like You Might Blackout (OHSA Item 1)
Description: OHSA item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug). All patients were on open-label droxidopa for 3 months prior to randomization to either continued droxidopa or to placebo.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 38 | 37
units on a scale | 0.9 (2.39) | 1.3 (2.21)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.251, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Patient Reported Clinical Global Impression - Severity
Description: The CGI-S is a 7 point scale ranging from a score of 1 (no symptoms) to 7 (severe symptoms). Patients were grouped according to OH severity at the end of the randomization period as follows;
  * Normal-Borderline OH (CGI-S 1-2),
  * Mild-Moderate OH (CGI-S 3-4),
  * Marked OH-Most Ill with OH (CGI-S 5-7). .
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 38 | 37
participants
  Normal-Borderline OH | 13 | 12
  Mild-Moderate OH | 16 | 13
  Marked OH-Most ill with OH | 9 | 12
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.708, Fisher Exact

7. Secondary Outcome: Clinician Recorded Clinical Global Impression - Severity
Description: The CGI-S is a 7 point scale ranging from a score of 1 (no symptoms) to 7 (severe symptoms). Patients were grouped according to OH severity at the end of the randomization period as follows;
  * Normal-Borderline OH (CGI-S 1-2),
  * Mild-Moderate OH (CGI-S 3-4),
  * Marked OH-Most Ill with OH (CGI-S 5-7).
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 38 | 37
participants
  Normal-Borderline OH | 9 | 7
  Mild-Moderate OH | 16 | 15
  Marked OH-Most ill with OH | 13 | 15
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.873, Fisher Exact

8. Secondary Outcome: Patient Reported Clinical Global Impression - Improvement
Description: The CGI-I is a 7 point scale ranging from a score of 1 (very much improved) to 7 (very much worse), with no change in the middle, and assesses the improvement in relation to the baseline evaluation.
  Patients will be grouped according change in disease as follows;
  * Very Much Improved to Slightly Improved (CGI-I 1-3),
  * No Change (CGI-I 4),
  * Slightly Worse to Very Much Worse (CGI-I 5-7).
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 38 | 37
participants
  Very much - Slightly Improved | 25 | 20
  No Change | 7 | 5
  Slightly - Very much Worse | 6 | 12
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.252, Fisher Exact

9. Secondary Outcome: Clinician Rated Clinical Global Impressions - Improvement
Description: as for outcome 8
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 38 | 37
participants
  Very much - Slightly Improved | 26 | 20
  No Change | 4 | 8
  Slightly - Very much Worse | 8 | 9
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.330, Fisher Exact

ADVERSE EVENTS:
Groups:
- Three Month Open-Label Droxidopa: all patients who participated in 3 months of open-label treatment with droxidopa (t.i.d., at optimal dose)
- Long-Term Follow-up: Open-label treatment with droxidopa (t.i.d) following the double-blind randomization phase.
- Total Droxidopa: All Patients exposed to droxidopa
Arm/Group | Three Month Open-Label Droxidopa | Double-blind Droxidopa | Double-blind Placebo | Long-Term Follow-up | Total Droxidopa
Serious Adverse Events (participants affected / at risk) | 12/102 | 1/38 | 0/37 | 16/74 | 26/102
Other Adverse Events (participants affected / at risk) | 37/102 | 8/38 | 4/37 | 43/74 | 62/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Three Month Open-Label Droxidopa (N=102) | Double-blind Droxidopa (N=38) | Double-blind Placebo (N=37) | Long-Term Follow-up (N=74) | Total Droxidopa (N=102)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Three Month Open-Label Droxidopa (N=102) | Double-blind Droxidopa (N=38) | Double-blind Placebo (N=37) | Long-Term Follow-up (N=74) | Total Droxidopa (N=102)
Headache (Nervous system disorders) | 5 (6) | 1 (1) | 2 (2) | 6 (6) | 13 (15)
Syncope (Nervous system disorders) | 4 (5) | 1 (2) | 0 (0) | 7 (9) | 10 (17)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (8) | 8 (12)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 5 (7)
Urinary Tract Infection (Infections and infestations) | 9 (10) | 2 (2) | 0 (0) | 11 (18) | 17 (31)
Bacteriuria (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 7 (8) | 11 (14)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 7 (8) | 0 (0) | 1 (1) | 16 (20) | 20 (29)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Orthostatic hypotension (Vascular disorders) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 6 (7)
Edema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (5)
Somnolence (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less